CLINICAL TRIAL: NCT05886166
Title: Clinical Utility of Exoskeleton Robot Training in Patients With Septic Arthritis After a Thermal Injury: A Case Report
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, So Young Joo, Hangang Sacred Heart Hospital IRB, Hangang Sacred Heart Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-16
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Septic Arthritis; Gait Disorder, Sensorimotor
MeSH Terms: conditions — Arthritis, Infectious; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Rebless® (H-ROBOTICS, KOREA) is a knee or ankle robot for range of motion (ROM) and strength training that can operate in passive or active mode in knee or ankle flexion and extension. The patients underwent 30 min of robot training using Rebless® with 30 min conventional therapy, 5 days a week for 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- robot assisted training (Experimental): Rebless® (H-ROBOTICS, KOREA) is a knee or ankle robot for range of motion (ROM) and strength training that can operate in passive or active mode in knee or ankle flexion and extension. The patients underwent 30 min of robot training using Rebless® with 30 min conventional therapy, 5 days a week for 8 weeks.
  Interventions: Other: robot assisted training

INTERVENTIONS:
Other: robot assisted training — Rebless® (H-ROBOTICS, KOREA) is a knee or ankle robot for range of motion (ROM) and strength training that can operate in passive or active mode in knee or ankle flexion and extension. The patients underwent 30 min of robot training using Rebless® with 30 min conventional therapy, 5 days a week for 8 weeks.

SUMMARY:
Bone and/or joint infections, such as septic arthritis (SA), are rare, but delayed diagnosis or improper treatment can result in irreversible joint destruction. Therefore, early diagnosis and effective treatment are necessary to prevent severe outcomes. Clear protocols for SA rehabilitation are unavailable, and physiotherapy studies are few. Robot training in patients with musculoskeletal diseases, including burns, can reduce pain and improve lower extremity function. Studies on robot training have been conducted in patients with burn injuries. Rebless® (H-ROBOTICS, KOREA) is a knee or ankle robot for range of motion (ROM) and strength training that can operate in passive or active mode in knee or ankle flexion and extension.

The patients underwent 30 min of robot training using Rebless® with 30 min conventional therapy, 5 days a week for 8 weeks.

This study aims to confirm the clinical effect after 8 weeks of robotic treatment for patients diagnosed with septic arthritis.

DETAILED DESCRIPTION:
Bone and/or joint infections, such as septic arthritis (SA), are rare, but delayed diagnosis or improper treatment can result in irreversible joint destruction. Therefore, early diagnosis and effective treatment are necessary to prevent severe outcomes. Clear protocols for SA rehabilitation are unavailable, and physiotherapy studies are few. Robot training in patients with musculoskeletal diseases, including burns, can reduce pain and improve lower extremity function. Studies on robot training have been conducted in patients with burn injuries. Rebless® (H-ROBOTICS, KOREA) is a knee or ankle robot for range of motion (ROM) and strength training that can operate in passive or active mode in knee or ankle flexion and extension.

Patients who underwent split thickness skin graft (STSG) at Hangang Sacred Heart Hospital, diagnosed with septic arthritis, aged >18 years, when weight bearing is not possible during intravenous antibiotic treatment in this study. This study excluded patients who had musculoskeletal diseases (fracture, amputation, rheumatoid arthritis, and degenerative joint diseases) involving the burned lower extremity. Patients with cognitive disorders, intellectual impairment before burn injury, serious cardiac dysfunction, problems with body weight ≥100 kg due to the belt length for fixing the thigh and calf, severe fixed contracture, skin disorders that could be worsened by RAGT, and severe pain who were unable to undergo rehabilitation programs were excluded.

The patients underwent 30 min of robot training using Rebless® with 30 min conventional therapy, 5 days a week for 8 weeks.

This study aims to confirm the clinical effect after 8 weeks of robotic treatment for patients diagnosed with septic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with septic arthritis
* aged >18 years, < 75 years
* when weight bearing is not possible during intravenous antibiotic treatment in this study.

Exclusion Criteria:

* had musculoskeletal diseases (fracture, amputation, rheumatoid arthritis, and degenerative joint diseases)
* cognitive disorders
* intellectual impairment before burn injury
* serious cardiac dysfunction
* skin disorders that could be worsened by robot training

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional ambulatory category (FAC) | 8 weeks
  6-point scale: 0, the patient could not walk or could only walk with the assistance of two people and 5, the patient can walk independently.

SECONDARY OUTCOMES:
6-min walking test (6 MWT) distance | 8 weeks
  6MWT measures the maximum distance a participant can walk in 6 min on a 20 m flat surface.
visual analog scale (VAS) | 8 weeks
  The visual analog scale (VAS) is used to assess subjective pain, with 0 representing no pain and 10 representing unbearable pain.
Isometric muscle strength | 8weeks
  Isometric muscle strength (hip, knee, and ankle) was measured using a microFET IITM (Hoggan Health Industries, Draper, UT, USA). Each trial lasted for 3-5 s, with a 30-s rest period between trials
range of motion (ROM) | 8 weeks
  The highest values obtained from the two valid measurements were recorded. The active ROMs of different joints (hip, knee, and ankle) were measured using a goniometer following a standardized technique.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Couderc M, Bart G, Coiffier G, Godot S, Seror R, Ziza JM, Coquerelle P, Darrieutort-Laffite C, Lormeau C, Salliot C, Veillard E, Bernard L, Baldeyrou M, Bauer T, Hyem B, Touitou R, Fouquet B, Mulleman D, Flipo RM, Guggenbuhl P; French Rheumatology Society Bone, Joint Infection Working Group. 2020 French recommendations on the management of septic arthritis in an adult native joint. Joint Bone Spine. 2020 Dec;87(6):538-547. doi: 10.1016/j.jbspin.2020.07.012. Epub 2020 Aug 3. PMID 32758534
- [Result] Barret JP, Desai MH, Herndon DN. Osteomyelitis in burn patients requiring skeletal fixation. Burns. 2000 Aug;26(5):487-9. doi: 10.1016/s0305-4179(99)00182-5. PMID 10812274
- [Result] Ju F, Wang Y, Xie B, Mi Y, Zhao M, Cao J. The Use of Sports Rehabilitation Robotics to Assist in the Recovery of Physical Abilities in Elderly Patients with Degenerative Diseases: A Literature Review. Healthcare (Basel). 2023 Jan 21;11(3):326. doi: 10.3390/healthcare11030326. PMID 36766901